CLINICAL TRIAL: NCT05733754
Title: Proteinuria as an Early Prognostic Factor for Detecting Possible Renal Affection After Liver Transplantation, a Single Egyptian Center Study
Brief Title: Proteinuria in Liver Transplantation, a Single Egyptian Center Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa M.Abokresha, principle investigator, Assiut University
Other Study IDs: Proteinuria
Record Dates: First submitted 2022-02-26; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Proteinuria has been suggested to be a predictive factor and an important tool for differentiating the etiology of renal dysfunction in various clinical scenarios .The good predictive performance of preoperative proteinuria utilized for the development of renal failure after operation has been reported . In the literature, prognostic significance of several scoring systems for end-stage liver disease has been validated . The Sequential Organ Failure Assessment (SOFA) system was found to be superior to ChildPugh points (CP points) and Model for End-Stage Liver Disease (MELD) score, and postoperative day 7 SOFA had the best discriminative power for predicting 3-month and 1-year mortality after liver transplantation . Renal dysfunction is one of the most significant adverse events in patients awaiting or undergoing a liver transplant, and its occurrence generally indicates a high rate of poor prognosis

DETAILED DESCRIPTION:
Proteinuria has been suggested to be a predictive factor and an important tool for differentiating the etiology of renal dysfunction in various clinical scenarios .The good predictive performance of preoperative proteinuria utilized for the development of renal failure after operation has been reported . In the literature, prognostic significance of several scoring systems for end-stage liver disease has been validated . The Sequential Organ Failure Assessment (SOFA) system was found to be superior to ChildPugh points (CP points) and Model for End-Stage Liver Disease (MELD) score, and postoperative day 7 SOFA had the best discriminative power for predicting 3-month and 1-year mortality after liver transplantation .Renal dysfunction is one of the most significant adverse events in patients awaiting or undergoing a liver transplant, and its occurrence generally indicates a high rate of poor prognosis .

In spite of the fact that proteinuria has been increasingly considered as a significant manifestation of acute or chronic renal disease , no study clarify the association between presence of proteinuria and prognosis of patients undergoing liver transplant.

The aim of the study

Primary objective:

Assess proteinuria as an early marker of renal dysfunction for liver transplant.

Secondary objective:

Defining different risk factors causing proteinuria.

Patients and methods

1. Study design Retrospective study
2. Inclusion criteria A total of 70 patients with end-stage liver disease received liver transplant will be included.
3. Exclusion criteria

   * Patients less than 18 years of age.
   * Patients with end-stage renal disease.

All data of patients will include :

* Demographic information, etiologies of primary liver disease, clinical parameters, lab investigations including CBC, urea, creatinine, liver enzymes, hepatitis viral markers, CMV infection, lipid profile, fasting and 2hours post prandial glucose level, anesthesia time, operation time, duration of hospitalization and ICU stay, and outcome.
* Associated medical conditions as diabetes mellitus, hypertension, dyslipidemia .
* The urinary analysis before transplantation and follow up for 6 months if proteinuria is present .
* types of immunosuppression taken.
* Occurrence of dialysis (temporary)
* Severity of liver disease will be assessed by CP points and MELD score Statistical analysis

  1. An excel sheet well be performed for data collection
  2. Clinical and laboratory data will be statistically analyzed

ELIGIBILITY:
Inclusion Criteria:

* A total of 70 patients with end-stage liver disease received liver transplant will be included.

Exclusion Criteria:

* Patients less than 18 years of age.
* Patients with end-stage renal disease.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All data of patients will include :
  * Demographic information, etiologies of primary liver disease, clinical parameters, lab investigations including CBC, urea, creatinine, liver enzymes, hepatitis viral markers, CMV infection, lipid profile, fasting and 2hours post prandial glucose level, anesthesia time, operation time, duration of hospitalization and ICU stay, and outcome.
  * Associated medical conditions as diabetes mellitus, hypertension, dyslipidemia .
  * The urinary analysis before transplantation and follow up for 6 months if proteinuria is present .
  * types of immunosuppression taken.
  * Occurrence of dialysis (temporary)
  * Severity of liver disease will be assessed by CP points and MELD score
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Assess incidence of proteinuria as an early marker of renal dysfunction for liver transplant. | Baseline
  Clarify the association between presence of proteinuria as an early marker of renal dysfunction for liver transplant and prognosis of patients undergoing liver transplant by measurement of serum creatinine clearance and albumin creatinine ratio in urine

CONTACTS AND LOCATIONS:
Overall Officials: marwa m abokrsha, MD, Principal Investigator — Lecturerer of internal medicine Gastroenterology and hepatology; Ramy A Hassan, Md, Study Chair — Assistant professor of surgery; Ahmed m Taha, MD, Study Chair — Assistant professor of surgery; Lobna A Ahmed, MD, Principal Investigator — Professor of internal medicine Gastroenterology and hepatology; Reem E Mahdy, MD, Principal Investigator — Consultant of internal medicine and hepatology
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Glassock RJ. Is the presence of microalbuminuria a relevant marker of kidney disease? Curr Hypertens Rep. 2010 Oct;12(5):364-8. doi: 10.1007/s11906-010-0133-3. PMID 20686930
- [Background] Heller F, Frischmann S, Grunbaum M, Zidek W, Westhoff TH. Urinary calprotectin and the distinction between prerenal and intrinsic acute kidney injury. Clin J Am Soc Nephrol. 2011 Oct;6(10):2347-55. doi: 10.2215/CJN.02490311. Epub 2011 Sep 1. PMID 21885792
- [Background] Huang TM, Wu VC, Young GH, Lin YF, Shiao CC, Wu PC, Li WY, Yu HY, Hu FC, Lin JW, Chen YS, Lin YH, Wang SS, Hsu RB, Chang FC, Chou NK, Chu TS, Yeh YC, Tsai PR, Huang JW, Lin SL, Chen YM, Ko WJ, Wu KD; National Taiwan University Hospital Study Group of Acute Renal Failure. Preoperative proteinuria predicts adverse renal outcomes after coronary artery bypass grafting. J Am Soc Nephrol. 2011 Jan;22(1):156-63. doi: 10.1681/ASN.2010050553. Epub 2010 Nov 29. PMID 21115618
- [Background] Wehler M, Kokoska J, Reulbach U, Hahn EG, Strauss R. Short-term prognosis in critically ill patients with cirrhosis assessed by prognostic scoring systems. Hepatology. 2001 Aug;34(2):255-61. doi: 10.1053/jhep.2001.26522. PMID 11481609
- [Background] Cholongitas E, Senzolo M, Patch D, Shaw S, Hui C, Burroughs AK. Review article: scoring systems for assessing prognosis in critically ill adult cirrhotics. Aliment Pharmacol Ther. 2006 Aug 1;24(3):453-64. doi: 10.1111/j.1365-2036.2006.02998.x. PMID 16886911
- [Background] Pan HC, Jenq CC, Tsai MH, Fan PC, Chang CH, Chang MY, Tian YC, Hung CC, Fang JT, Yang CW, Chen YC. Scoring systems for 6-month mortality in critically ill cirrhotic patients: a prospective analysis of chronic liver failure - sequential organ failure assessment score (CLIF-SOFA). Aliment Pharmacol Ther. 2014 Nov;40(9):1056-65. doi: 10.1111/apt.12953. Epub 2014 Sep 11. PMID 25208465
- [Background] Wong CS, Lee WC, Jenq CC, Tian YC, Chang MY, Lin CY, Fang JT, Yang CW, Tsai MH, Shih HC, Chen YC. Scoring short-term mortality after liver transplantation. Liver Transpl. 2010 Feb;16(2):138-46. doi: 10.1002/lt.21969. PMID 20104481